CLINICAL TRIAL: NCT02344680
Title: Liver Fibrosis in Zambian HIV-HBV Co-infected Patients: a Long-term Prospective Cohort Study
Brief Title: Liver Fibrosis in Zambian HIV-HBV Co-infected Patients
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Michael Vinikoor, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: IRB-3000; K01TW009998 (NIH)
Record Dates: First submitted 2015-01-12; First posted 2015-01-26 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Human Immunodeficiency Virus; HBV; Fibrosis, Liver; Cirrhosis, Liver; Hepatocellular Carcinoma; Hepatitis Delta Virus; Alcoholic Hepatitis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Liver Cirrhosis; Carcinoma, Hepatocellular; Hepatitis D; Hepatitis, Alcoholic | interventions — Anti-HIV Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Adults with HIV-HBV co-infection: Adults with HIV-HBV co-infection who are receiving antiretroviral therapy
  Interventions: Drug: Anti-HIV Agents

INTERVENTIONS:
Drug: Anti-HIV Agents
  Other Names: Anti-retroviral therapy

SUMMARY:
A cohort of adults with HIV-HBV co-infection will be created in Lusaka, Zambia, to describe the short and long-term (up to 10 years of follow-up) HBV and liver outcomes, including the effectiveness of current therapies, and to identify the risk factors for major endpoints of interest, including HCC and HBV functional cure. This cohort will also create a pool of potential participants for in-depth mechanistic studies and clinical trials of novel HBV cure drugs.

DETAILED DESCRIPTION:
Among people with HIV in Africa, liver disease is a neglected area of investigation but is anticipated to become increasingly common as patients live longer due to antiretroviral therapy. In Lusaka, Zambia, we previously (NCT02060162, clinicaltrials.gov) described that HIV-HBV co-infection was the most important liver risk factor. However, in that study, only very short-term outcomes could be assessed. Building on these preliminary results and addressing the need to study HIV-HBV during a longer duration of follow-up, the current protocol will focus exclusively on people with HIV-HBV in Zambia. Zambia is an ideal site for this research as it has ~12% HIV prevalence and 6% HBsAg-positivity among adults nationwide. In fact, ~70% of people with HIV-HBV globally reside in Africa. In the proposed study, we will obtain consent from people with HIV-HBV to participate in an observational cohort study with up to 10 years of follow-up. Standard of care antiviral therapies will be received by participants. More in-depth analysis of liver and HBV viral and serological outcomes will occur. Screening for liver cancer will also occur. This study will provide useful clinical and epidemiological information to health policymakers in Zambia and beyond. It will also provide a platform for the training of health workers in Zambia in HBV clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Living with HIV infection
* Living with active HBV infection, defined as any single positive HBsAg assay
* Naïve to antiretroviral therapy or currently participating in HIV/HBV co-infection in IeDEA-SA

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Planning to relocate out of Lusaka district

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 adults with HIV-HBV coinfection
Sampling Method: Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in liver fibrosis stage | From baseline to 10 years of follow-up
  Measure of liver fibrosis using AST-to-platelet ratio index (APRI), Fibrosis 4 (FIB-4) and transient elastography. Ascertainment of potential risk factors including demographics, alcohol use, HIV-related biomarkers, HBV DNA, hepatitis delta virus, and other factors.

SECONDARY OUTCOMES:
Incidence of hepatocellular carcinoma | From baseline to 10 years of follow-up
  Number of new cases of hepatocellular carcinoma during follow-up
Prevalence of significant liver fibrosis (Metavir F2 or greater) | At enrollment
  Proportion of participants with liver fibrosis by non-invasive measures (AST-to-platelet ratio index, Fibrosis 4, or transient elastography)
Prevalence of persistent HBV viremia: Measure HBV DNA at month 24 | Month 24
  Proportion of participants with measure of HBV DNA above detection at month 24

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Vinikoor, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Centre for Infectious Disease Research in Zambia (CIDRZ), Lusaka, Lusaka Province, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weber R, Sabin CA, Friis-Moller N, Reiss P, El-Sadr WM, Kirk O, Dabis F, Law MG, Pradier C, De Wit S, Akerlund B, Calvo G, Monforte Ad, Rickenbach M, Ledergerber B, Phillips AN, Lundgren JD. Liver-related deaths in persons infected with the human immunodeficiency virus: the D:A:D study. Arch Intern Med. 2006 Aug 14-28;166(15):1632-41. doi: 10.1001/archinte.166.15.1632. PMID 16908797
- [Background] Central Statistical Office (CSO) MoH, Tropical Diseases Research Centre, University of Zambia, and Macro International Inc. Zambia Demographic and Health Survey 2007. Calverton, Maryland, USA: CSO and Macro International Inc., 2009.
- [Background] Kapembwa KC, Goldman JD, Lakhi S, Banda Y, Bowa K, Vermund SH, Mulenga J, Chama D, Chi BH. HIV, Hepatitis B, and Hepatitis C in Zambia. J Glob Infect Dis. 2011 Jul;3(3):269-74. doi: 10.4103/0974-777X.83534. PMID 21887060
- [Background] Hamers RL, Zaaijer HL, Wallis CL, Siwale M, Ive P, Botes ME, Sigaloff KC, Hoepelman AI, Stevens WS, Rinke de Wit TF; PharmAccess African Studies to Evaluate Resistance (PASER). HIV-HBV coinfection in Southern Africa and the effect of lamivudine- versus tenofovir-containing cART on HBV outcomes. J Acquir Immune Defic Syndr. 2013 Oct 1;64(2):174-82. doi: 10.1097/QAI.0b013e3182a60f7d. PMID 23892239
- [Background] Martin-Carbonero L, Teixeira T, Poveda E, Plaza Z, Vispo E, Gonzalez-Lahoz J, Soriano V. Clinical and virological outcomes in HIV-infected patients with chronic hepatitis B on long-term nucleos(t)ide analogues. AIDS. 2011 Jan 2;25(1):73-9. doi: 10.1097/QAD.0b013e328340fde2. PMID 21076274
- [Background] Tuma P, Medrano J, Resino S, Vispo E, Madejon A, Sanchez-Piedra C, Rivas P, Labarga P, Martin-Carbonero L, Barreiro P, Soriano V. Incidence of liver cirrhosis in HIV-infected patients with chronic hepatitis B or C in the era of highly active antiretroviral therapy. Antivir Ther. 2010;15(6):881-6. doi: 10.3851/IMP1630. PMID 20834100
- [Background] Kirk GD, Bah E, Montesano R. Molecular epidemiology of human liver cancer: insights into etiology, pathogenesis and prevention from The Gambia, West Africa. Carcinogenesis. 2006 Oct;27(10):2070-82. doi: 10.1093/carcin/bgl060. Epub 2006 May 5. PMID 16679307
- [Background] Stabinski L, Reynolds SJ, Ocama P, Laeyendecker O, Ndyanabo A, Kiggundu V, Boaz I, Gray RH, Wawer M, Thio C, Thomas DL, Quinn TC, Kirk GD; Rakai Health Sciences Program. High prevalence of liver fibrosis associated with HIV infection: a study in rural Rakai, Uganda. Antivir Ther. 2011;16(3):405-11. doi: 10.3851/IMP1783. PMID 21555823
- [Background] Crane M, Iser D, Lewin SR. Human immunodeficiency virus infection and the liver. World J Hepatol. 2012 Mar 27;4(3):91-8. doi: 10.4254/wjh.v4.i3.91. PMID 22489261
- [Background] Puoti M, Manno D, Nasta P, Carosi G. Hepatitis B virus and HIV coinfection in low-income countries: unmet needs. Clin Infect Dis. 2008 Feb 1;46(3):367-9. doi: 10.1086/525532. No abstract available. PMID 18171305
- [Background] Hoffmann CJ, Charalambous S, Martin DJ, Innes C, Churchyard GJ, Chaisson RE, Grant AD, Fielding KL, Thio CL. Hepatitis B virus infection and response to antiretroviral therapy (ART) in a South African ART program. Clin Infect Dis. 2008 Dec 1;47(11):1479-85. doi: 10.1086/593104. PMID 18937580
- [Background] Hawkins C, Christian B, Ye J, Nagu T, Aris E, Chalamilla G, Spiegelman D, Mugusi F, Mehta S, Fawzi W. Prevalence of hepatitis B co-infection and response to antiretroviral therapy among HIV-infected patients in Tanzania. AIDS. 2013 Mar 27;27(6):919-927. doi: 10.1097/QAD.0b013e32835cb9c8. PMID 23196935
- [Background] Wandeler G, Gsponer T, Bihl F, Bernasconi E, Cavassini M, Kovari H, Schmid P, Battegay M, Calmy A, Egger M, Furrer H, Rauch A; Swiss HIV Cohort Study. Hepatitis B virus infection is associated with impaired immunological recovery during antiretroviral therapy in the Swiss HIV cohort study. J Infect Dis. 2013 Nov 1;208(9):1454-8. doi: 10.1093/infdis/jit351. Epub 2013 Jul 30. PMID 23901088
- [Background] Easterbrook P, Sands A, Harmanci H. Challenges and priorities in the management of HIV/HBV and HIV/HCV coinfection in resource-limited settings. Semin Liver Dis. 2012 May;32(2):147-57. doi: 10.1055/s-0032-1316476. Epub 2012 Jul 3. PMID 22760654
- [Background] Kelly P, Saloojee H, Chen JY, Chung RT. Noncommunicable diseases in HIV infection in low- and middle-income countries: gastrointestinal, hepatic, and nutritional aspects. J Acquir Immune Defic Syndr. 2014 Sep 1;67 Suppl 1(0 1):S79-86. doi: 10.1097/QAI.0000000000000260. PMID 25117963
- [Background] Fattovich G, Bortolotti F, Donato F. Natural history of chronic hepatitis B: special emphasis on disease progression and prognostic factors. J Hepatol. 2008 Feb;48(2):335-52. doi: 10.1016/j.jhep.2007.11.011. Epub 2007 Dec 4. PMID 18096267
- [Background] Puoti M, Torti C, Bruno R, Filice G, Carosi G. Natural history of chronic hepatitis B in co-infected patients. J Hepatol. 2006;44(1 Suppl):S65-70. doi: 10.1016/j.jhep.2005.11.015. Epub 2005 Nov 28. PMID 16338021
- [Background] Thio CL. Hepatitis B in the human immunodeficiency virus-infected patient: epidemiology, natural history, and treatment. Semin Liver Dis. 2003 May;23(2):125-36. doi: 10.1055/s-2003-39951. PMID 12800066
- [Background] Lok AS. Chronic hepatitis B. N Engl J Med. 2002 May 30;346(22):1682-3. doi: 10.1056/NEJM200205303462202. No abstract available. PMID 12037146
- [Background] Hoffmann CJ, Thio CL. Clinical implications of HIV and hepatitis B co-infection in Asia and Africa. Lancet Infect Dis. 2007 Jun;7(6):402-9. doi: 10.1016/S1473-3099(07)70135-4. PMID 17521593
- [Background] Thio CL, Seaberg EC, Skolasky R Jr, Phair J, Visscher B, Munoz A, Thomas DL; Multicenter AIDS Cohort Study. HIV-1, hepatitis B virus, and risk of liver-related mortality in the Multicenter Cohort Study (MACS). Lancet. 2002 Dec 14;360(9349):1921-6. doi: 10.1016/s0140-6736(02)11913-1. PMID 12493258
- [Background] Zambian Ministry of Health. Guidelines for the care of individuals with HIV/AIDS, 2010.
- [Background] Consolidated Guidelines on the Use of Antiretroviral Drugs for Treating and Preventing HIV Infection: Recommendations for a Public Health Approach. Geneva: World Health Organization; 2013 Jun. Available from http://www.ncbi.nlm.nih.gov/books/NBK195400/ PMID 24716260
- [Background] Sterling RK, Lissen E, Clumeck N, Sola R, Correa MC, Montaner J, S Sulkowski M, Torriani FJ, Dieterich DT, Thomas DL, Messinger D, Nelson M; APRICOT Clinical Investigators. Development of a simple noninvasive index to predict significant fibrosis in patients with HIV/HCV coinfection. Hepatology. 2006 Jun;43(6):1317-25. doi: 10.1002/hep.21178. PMID 16729309
- [Background] Wai CT, Greenson JK, Fontana RJ, Kalbfleisch JD, Marrero JA, Conjeevaram HS, Lok AS. A simple noninvasive index can predict both significant fibrosis and cirrhosis in patients with chronic hepatitis C. Hepatology. 2003 Aug;38(2):518-26. doi: 10.1053/jhep.2003.50346. PMID 12883497
- [Background] Sandrin L, Fourquet B, Hasquenoph JM, Yon S, Fournier C, Mal F, Christidis C, Ziol M, Poulet B, Kazemi F, Beaugrand M, Palau R. Transient elastography: a new noninvasive method for assessment of hepatic fibrosis. Ultrasound Med Biol. 2003 Dec;29(12):1705-13. doi: 10.1016/j.ultrasmedbio.2003.07.001. PMID 14698338
- [Background] Hawkins C, Agbaji O, Ugoagwu P, Thio CL, Auwal MM, Ani C, Okafo C, Wallender E, Murphy RL. Assessment of liver fibrosis by transient elastography in patients with HIV and hepatitis B virus coinfection in Nigeria. Clin Infect Dis. 2013 Dec;57(12):e189-92. doi: 10.1093/cid/cit564. Epub 2013 Sep 6. PMID 24014732
- [Background] Bonnard P, Sombie R, Lescure FX, Bougouma A, Guiard-Schmid JB, Poynard T, Cales P, Housset C, Callard P, Le Pendeven C, Drabo J, Carrat F, Pialoux G. Comparison of elastography, serum marker scores, and histology for the assessment of liver fibrosis in hepatitis B virus (HBV)-infected patients in Burkina Faso. Am J Trop Med Hyg. 2010 Mar;82(3):454-8. doi: 10.4269/ajtmh.2010.09-0088. PMID 20207872
- [Background] Marcellin P, Gane E, Buti M, Afdhal N, Sievert W, Jacobson IM, Washington MK, Germanidis G, Flaherty JF, Aguilar Schall R, Bornstein JD, Kitrinos KM, Subramanian GM, McHutchison JG, Heathcote EJ. Regression of cirrhosis during treatment with tenofovir disoproxil fumarate for chronic hepatitis B: a 5-year open-label follow-up study. Lancet. 2013 Feb 9;381(9865):468-75. doi: 10.1016/S0140-6736(12)61425-1. Epub 2012 Dec 10. PMID 23234725
- [Background] Cardoso AC, Carvalho-Filho RJ, Stern C, Dipumpo A, Giuily N, Ripault MP, Asselah T, Boyer N, Lada O, Castelnau C, Martinot-Peignoux M, Valla DC, Bedossa P, Marcellin P. Direct comparison of diagnostic performance of transient elastography in patients with chronic hepatitis B and chronic hepatitis C. Liver Int. 2012 Apr;32(4):612-21. doi: 10.1111/j.1478-3231.2011.02660.x. Epub 2011 Nov 22. PMID 22103765
- [Background] Miailhes P, Pradat P, Chevallier M, Lacombe K, Bailly F, Cotte L, Trabaud MA, Boibieux A, Bottero J, Trepo C, Zoulim F. Proficiency of transient elastography compared to liver biopsy for the assessment of fibrosis in HIV/HBV-coinfected patients. J Viral Hepat. 2011 Jan;18(1):61-9. doi: 10.1111/j.1365-2893.2010.01275.x. PMID 20196798
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Vinikoor MJ, Schuttner L, Moyo C, Li M, Musonda P, Hachaambwa LM, Stringer JS, Chi BH. Short communication: Late refills during the first year of antiretroviral therapy predict mortality and program failure among HIV-infected adults in urban Zambia. AIDS Res Hum Retroviruses. 2014 Jan;30(1):74-7. doi: 10.1089/AID.2013.0167. Epub 2013 Aug 30. PMID 23924188
- [Background] Kim BK, Fung J, Yuen MF, Kim SU. Clinical application of liver stiffness measurement using transient elastography in chronic liver disease from longitudinal perspectives. World J Gastroenterol. 2013 Mar 28;19(12):1890-900. doi: 10.3748/wjg.v19.i12.1890. PMID 23569334
- [Background] The Zambian National Health Research Bill, 2013